CLINICAL TRIAL: NCT03205267
Title: Multicenter, Open-label Single Arm Phase II Study Testing the Tolerability and the Efficacy of Bosutinib step-in Dosing in Chronic Phase CML Patients Intolerant or Refractory to Previous Imatinib, Nilotinib or Dasatinib Therapy
Brief Title: Phase II Study Testing the Tolerability and the Efficacy of Bosutinib in Chronic Phase CML Patients
Acronym: BODO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bonn (Other)
Collaborators: RWTH Aachen University (Other); Ludwig-Maximilians - University of Munich (Other); University of Jena (Other); Heidelberg University (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Dominik Wolf, Principal Investigator Prof. Dr. med. D. Wolf, University of Bonn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED3-201401-BODO; 2014-005531-13 (EudraCT Number)
Record Dates: First submitted 2017-05-29; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Chronic Myelogenous Leukaemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bosutinib (Experimental): Drug: Bosulif 100 mg or 500 mg tablets step in dosing scheme
  Interventions: Drug: Bosulif

INTERVENTIONS:
Drug: Bosulif — Patients will start with dose-level 1 (300 mg once daily) Bosutinib. If patients do not experience any toxicity or only G1 toxicity, they will be dose-increased first to dose-level 2 (400 mg once daily ) and then to dose-level 3 (500 mg once daily). Dose will not be escalated above 500 mg which is the dose recommended by the summary of product information. If patients experience G2 toxicity, the study drug will be further continued at the same dose-level. In patients with G3 or G4 toxicities, therapy will be withheld until toxicity resolved to <G2.
  Other Names: Bosutinib

SUMMARY:
Bosutinib is a 2nd generation tyrosine kinase inhibitor that has shown promising results from first up to fourth line treatment in patients with in chronic phase of chronic myelogenous leukaemia. Most patients discontinuing the treatment with Bosutinib do so because of side effects occuring early after starting the treatment. A step in dosing scheme could improve these early toxicities. The aim of this study therefore is to demonstrate that temporary lowering of the Bosutinib dose during early treatment may help to reduce or prevent side effects while preserving efficacy.

DETAILED DESCRIPTION:
Objectives:

The objective of the BODO trial is to assess the tolerability and efficacy of a step-in dosing concept of the dual SRC-ABL kinase inhibitor Bosutinib in CP-CML patients who either developed intolerance or treatment failure to previous Imatinib, Dasatinib or Nilotinib as 1st line therapy.

Primary endpoint:

• Rate of GI-Toxicity (i.e. incidence and severity of grade 2 to 4 toxicities) within the first 6 months of treatment

Secondary endpoints:

* Tolerability (i.e. all grade, grade 2 to 4 and grade 3 and 4 toxicities) at month 6, 12 and 24
* Efficacy parameters: CCyR, MMR, MR4 and MR4.5 rate at month 3, 6, 12, 18 and 24
* Patient-reported outcome measures (QoL)
* Progression-free survival (PFS)
* Overall survival (OS)
* The rate of emerging mutations during Bosutinib treatment

Exploratory endpoints linked to substudies:

Vascular biology substudy:

* Effects of previous therapy on the baseline vascular risk profile (i.e. Nilotinib- vs. Dasatinib-pre-treatment)
* Biological and clinical surrogates for vascular alterations during Bosutinib therapy at baseline, months 6, 12, and 24

Pharmacokinetic (PK), pharmacodynamic (PD) and immunology sub- study:

* Correlation of PK with response and toxicity
* Correlation of PK with PD (i.e. phosphoproteomic changes) in immune cell populations
* Correlation of PD changes in immune cell populations with response
* Evaluation of the effects of Bosutinib on frequency and phenotype of immune cells
* Evaluation whether Bosutinib-induced changes of immune cells correlate to response

Ultra-deep next-generation sequencing (UD-NGS) and telomere substudy:

* Documentation of subclone evolution or elimination during Bosutinib treatment
* Evaluation of telomere length in leukemic and non-leukemic cells as a prognostic indicator for depth and kinetics of response to and tolerability of Bosutinib

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female patients aged ≥18 years
* ECOG performance status of 0 to 2
* CML in 1st or late chronic phase
* Intolerant or resistant to pretreatment with one of the approved 1st line TKIs (Imatinib, Nilotinib or Dasatinib). Imatinib therapy prior to 2nd generation TKI therapy for a maximum of 6 weeks is allowed.
* Patients must have a serum creatinine of ≤ 2 x ULN, SGOT/SGPT ≤ 3 x ULN, total bilirubin ≤ 2 x ULN (except known Gilbert's syndrome), and Lipase ≤ 1.5 x ULN
* Female patients of childbearing potential must have a negative pregnancy test performed during screening period
* Male and female patients of reproductive potential must currently use a highly effective contraceptive method and be willing to keep on using it throughout the study and for 6 months following discontinuation of study drug.

Exclusion Criteria:

* Hypersensitivity against Bosutinib or other ingredients of the medicinal product
* Evidence of features of accelerated (AP) or blast phase (BC) at any time before inclusion
* Patients with BCR-ABL negative CML
* Patients having received Imatinib for more than 6 weeks prior to initiation of 2nd generation TKI (either Nilotinib or Dasatinib)
* Patients with known T315I or V299L mutation
* Concomitant medications known to be strong inducers or inhibitors of P450 isoenzyme CYP3A4
* History of pancreatitis, inflammatory bowel disease requiring systemic or topical immunosuppressive therapy within the last 12 months
* Impaired cardiac function, including any of the following:

  1. History of or presence of complete left bundle branch block, right bundle branch block plus left anterior hemiblock, bifascicular block in screening ECG
  2. ST depression of >1mm in 2 or more leads and/or T wave inversions in 2 or more contiguous leads in screening ECG
  3. Congenital long QT syndrome
  4. QTc> 450 msec in the screening ECG
  5. QT-prolonging concomitant medication
  6. History of or presence of significant ventricular or atrial tachyarrhythmias in screening ECG
  7. History of or presence of clinically significant resting bradycardia (< 50 beats per minute)
  8. Myocardial infarction within 6 months prior to inclusion
  9. Unstable angina diagnosed or treated during the past 12 months
  10. Uncontrolled hypertension, history of labile hypertension
* Known HIV and/or active viral hepatitis (hepatitis B or C). Hepatitis B screening will be performed at screening. Patients with history of hepatitis B with negative HBV DNA may be included when using antiviral prophylaxis
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinoma of the skin
* Treatment with another investigational product during this study or during the last 30 days prior to study start, except treatment with Interferon alpha within the TIGER (CML V) protocol, which must be stopped at least 7 days prior to study entry
* Any circumstance at the time of study entry that would preclude completion of the study or the required follow-up prohibits inclusion into this study
* Patient must not have any active bacterial, viral or fungal infection at screening
* Patient must not have severe cerebral dysfunction and/or legal incapacity
* Conditions which interfere with the study treatment at the discretion of the investigator
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Rate of GI-Toxicity (i.e. incidence and severity of grade 2 to 4 toxicities) | within the first 6 months of treatment
  calculation of the incidence rate of grade 2 to 4 GI toxicity with and without regard to causality

SECONDARY OUTCOMES:
overall Tolerability (i.e. all grade, grade 2 to 4 and grade 3 and 4 toxicities) | at month 6, 12 and 24
  Apart from grade 2 to 4 GI toxicity, the occurrence of toxicity will be analyzed in general. This regards all grade toxicity, 2 to 4 grade and 3 to 4 grade toxicity (NCI CTCAE v4.0).
Molecular response mesured by efficacy parametern | at month 3, 6, 12, 18 and 24
  Rating of CCyR, MMR, MR4 and MR4.5 after bone marrow aspiration and biopsy
Patient-reported outcome measures (QoL) | at month 3 and 6
  The EORTC QLQ-CML30 will be scored according to the respective user's guides.
Progression-free survival (PFS) | at month 3, 6, 9, 12, 15, 18, 21 and 24
  Progression will be assessed according to the visit schedule at any visit.
Overall Survival (OS) | at month 3, 6, 9, 12, 15, 18, 21 and 24
  Survival will be assessed according to the visit schedule at any visit.
The rate of emerging mutations during Bosutinib treatment | at month 3, 6, 9, 12, 15, 18, 21 and 24
  The rate and type of mutations will be described. The rate will be given as percentage of patients developing mutations.

OTHER OUTCOMES:
Vascular biology substudy: analysis of clinical and laboratory vascular and metabolic risk factors | baseline, at months 6, 12 and 24
  Ankle Brachial Index (ABI) will be prospectively evaluated followed by analysis of various biomarkers for vascular damage
Pharmacokinetic (PK), pharmacodynamic (PD) substudy | at day 1, months 1, 2, 3, 12, 18, 24
  It is planned to analyze PK parameters sequentially by taking serum from PB and subsequent HPLC-MS/MS technology. Pharmacodynamics in different compartments will be analyzed by means of flow-cytometry of PB and BM samples.
Telomere substudy | at months 1, 2, 3, 12 and 24
  Assessment of telomere length in normal and leukemic cells as potential new biomarker for prognosis, prediction of response under Bosutinib
Ultra-deep next-generation sequencing (UD-NGS) | at months 1, 2, 3, 12 and 24
  Documentation of subclone evolution or elimination during Bosutinib treatment
Assessment of patients comorbidities and correlation to individual patient´s adverse side effect profile substudy | through study completion, an average of 2 years
  Documentation of patient´s comorbidity profile using 3 different comorbidity scales
Transport mechanisms of Bosutinib and mechanisms of diarrhea substudy | every 14 days month 1-3
  Investigation the role of the 5-HT pathway in directing bosutinib induced diarrhea by assessment of 5-HT and certain cytokine levels and genetic analysis including SNP and GWAS

CONTACTS AND LOCATIONS:
Overall Officials: Dominik GF Wolf, Prof. Dr., Principal Investigator — University of Bonn Medical Faculty; Brümmendorf H Tim, Prof. Dr., Study Chair — University of Aachen Medical Faculty
Locations (1):
- University Hospital Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No